CLINICAL TRIAL: NCT02370758
Title: Cell Mediated Immunity as a Guide for Secondary Prophylaxis in SOT Patients With CMV Infection
Brief Title: Cell Mediated Immunity for Secondary Prophylaxis in CMV SOT Patients
Acronym: Q-CMV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UHN-CMV-001
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Cytomegalovirus Viraemia
Keywords: Quantiferon-CMV; Quantiferon-Monitor; Solid Organ Transplants; CMV Disease
MeSH Terms: interventions — Valganciclovir; Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low CMV CMI (Active Comparator): Patients that show low levels of cell-mediated immunity against CMV will have their antiviral therapy (oral Valganciclovir or Intravenous Ganciclovir) continued for an additional 2 months at half dose.
  Interventions: Drug: Valganciclovir or Ganciclovir
- High CMV CMI (No Intervention): Patients that show high levels of cell-mediated immunity against CMV will have their antiviral therapy (oral Valganciclovir or Intravenous Ganciclovir) stopped.

INTERVENTIONS:
Drug: Valganciclovir or Ganciclovir
  Arms: Low CMV CMI

SUMMARY:
This study will evaluate whether a test for Cytomegalovirus (CMV) specific cell-mediated immunity can be used to determine whether patients who complete a course of therapy for CMV viremia need secondary antiviral prophylaxis. Subjects that have negative CMV CMI will receive antiviral prophylaxis for 2 months and those with positive CMV CMI will have their prophylaxis stopped.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) is the most important infection in transplant patients and it is a common cause of illness in patients who have undergone a transplant. Serious infections due to CMV can affect many parts of the body including the lungs, the gut, and the liver; when CMV infection becomes serious enough to cause symptoms, it is called CMV disease. Some patients require treatment while others will clear the virus on their own.

QuantiFERON-CMV (QFT-CMV) is a blood test that measures CMV-specific cell-mediated immunity. This test was able to predict that patients with low cell-mediated immunity are at greater risk for developing CMV disease. In this study, QFT-CMV will be used to make a decision regarding CMV treatment. The QFT-CMV test will be performed at the first detection of CMV, at end of antiviral therapy and one month post-therapy. The end-of-therapy results will be available to clinicians and study investigators within one week of collection. Based on the result, a decision will be made to continue with prolonged antiviral therapy. Patients that show weak cell-mediated immunity against CMV will be given secondary antiviral prophylaxis, while patients with good cell-mediated immunity will have their therapy stopped. Patients will continue to be monitored three months after the last QFT-CMV test for recurrent CMV viremia.

This study will also attempt to evaluate the predictive value of the QuantiFERON-Monitor (QFT-Monitor) assay. QFT-Monitor is a recently developed non-pathogen specific immune assay: it is based on immune activation of both innate and adaptive immunity. The investigators hypothesize that stimulation of both the innate and adaptive immunity may predict global immune function and also be predictive of CMV reactivation. The investigators plan to perform the QFT-Monitor assay in parallel to the QFT-CMV test to determine the test characteristics and cut-off values in predicting global immune function. This test will be collected and tested in batches. Therefore, the results will not influence clinical decisions.

ELIGIBILITY:
Inclusion Criteria:

* Adult solid organ transplant (SOT) recipient on at least one immunosuppressive medication
* Starting therapy for new onset asymptomatic CMV viremia OR starting therapy for new onset CMV disease
* CMV viral load ≥ 1000 IU/mL

Exclusion Criteria:

* Known ganciclovir-resistant CMV
* Known intolerance to valganciclovir or ganciclovir
* Unable to comply with protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Virologic recurrence or disease recurrence | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Atul Humar, MD, Principal Investigator — University Health Network, Toronto; Deepali Kumar, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto General Hospital, Multi-Organ Transplant, Toronto, Ontario, Canada